CLINICAL TRIAL: NCT03442179
Title: Cognitive Outcomes and Neuroimages Associated With Anesthesia-Related EEG Signatures
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patrick L. Purdon, Associate Professor of Anaesthesia, Massachusetts General Hospital
Other Study IDs: 2017P000413
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Elderly; General Anesthesia
Keywords: Aging; Anesthesia; EEG monitoring; Burst suppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to assess inflammatory markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we propose to evaluate the relationship between the alpha oscillation dynamics and the signals derived from the brain images related to brain aging.

DETAILED DESCRIPTION:
In 1955 Bedford reported the "adverse cerebral effects of anesthesia on old people" and suggested precautions in relation to operations on the elderly. Since then, many studies have investigated the incidence of and the risk factors for postoperative cognitive dysfunction (POCD). The incidence ranges from 8.9% to 46.1% and advanced age, preoperative mild cognitive impairment, extensive surgical procedures and other factors have been identified as important risk factors. The incidence has been reported to be as high as 41.4% at hospital discharge and 12.7% at 3 months after surgery in the elderly (60 years or older). Postoperative delirium (POD) is a more acute complication of major surgery, affecting 10-70% of surgical patients 60 years and older. Some studies have shown the association between POD and early POCD, and even POD and POCD are commonly reported as being part of the same continuum. Whether this is true or not, both represent postoperative cognitive deterioration, and age is the predominant risk factor for both.

Every day in the United States, nearly 100,000 patients undergo general anesthesia and sedation for surgical and diagnostic procedures. Approximately 35% of all surgical procedures are performed on adults older than 65 years. Considering the aging surgical population, the burden of postoperative cognitive disorders will almost certainly increase over time.

Although many factors, such as surgical stress, inflammation, and other comorbidities may contribute to POCD, there is evidence that anesthetic exposure plays a major role. Pre-clinical studies have demonstrated that exposure to anesthetic drugs is neurotoxic, and that older animals are particularly vulnerable. It is also generally understood that the elderly are more sensitive to anesthetics, meaning that lower doses of anesthetic drugs are required to induce and maintain unconsciousness. This has led to age-adjusted guidelines for anesthetic dosing, which in theory could be used to mitigate potentially harmful anesthetic exposures. However, these guidelines describe the age-dependent dose-response relationships for a population of patients; individual drug requirements can vary significantly, by a factor of ~2 above or below the levels recommended by population-based models. In the absence of a means to measure and monitor individual drug responses, anesthesiologists would tend to err on the side of administering more anesthetic than required, to minimize the probability of patient awareness across the population as a whole.

Fortunately, in recent years, significant progress has been made to understand the neural mechanisms of anesthesia-induced unconsciousness, making it possible to monitor individual patients' drug responses using the electroencephalogram (EEG). Increasing concentrations of the commonly-used GABAergic anesthetic drugs, such as propofol and sevoflurane, induce a stereotyped sequence of brain oscillations with increasing drug concentration. These brain oscillations are directly related to the states of sedation and unconsciousness induced by anesthetic drugs, and readily observed using the EEG. At lower concentrations, propofol and sevoflurane, two of the most commonly used anesthetic drugs, induce beta oscillations (12-25 Hz). At concentrations producing unconsciousness for general anesthesia, these drugs produce frontal alpha (8-12 Hz) and slow (0.1 to 1 Hz) oscillations. At still higher concentrations, propofol and sevoflurane produce a pattern referred to as burst suppression, a deep state of brain inactivation in which brain activity is punctuated by long periods of neuronal and EEG silence. However, it is now known that elderly patients do not always exhibit this canonical EEG signature under general anesthesia. First, it was described that ageing was associated with a decrease in the frontal alpha power. Then, other studies suggested that older patients with poor preoperative cognitive performance also lack the alpha band under anesthesia. And finally, our group demonstrated that a low alpha power is also associated with a higher risk to develop burst suppression under anesthesia. Nonetheless, the potential mechanism related to the lower alpha power with ageing and cognitive function remains unknown. In this study, we propose to evaluate the relationship between the alpha oscillation dynamics and the signals derived from brain images related to brain aging.

We hypothesize that: 1) Brain imaging signals will correlate with the alpha power induced by anesthetics, and 2) Aging brain imaging features will be associated with postoperative cognitive recovery.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or above (male and female)
* American Society of Anesthesiologists (ASA) physical status classification of I, II or III.
* Candidates scheduled for open or laparoscopic general surgical procedures under general anesthesia
* No cognitive impairment base on Telephone Interview for Cognitive Status (TICS)
* Fluency in English Language

Exclusion Criteria:

* Prior diagnosis of dementia
* Prior diagnosis of Alzheimer's Disease
* Prior history of psychiatric or neurological diseases including:
* Schizophrenia
* Parkinsonism
* Epilepsy or seizure
* Brain injury
* Brain tumors/metastases
* Encephalitis
* Stroke, CVA, TIA
* Drug or alcohol abuse:
* Any history of IV drug abuse
* Alcohol/drug (non-IV) abuse <10 years
* Language impairment
* Hearing or visual impairment
* Severe obesity (BMI ≥40 kg/m2)
* MRI contraindications, such as presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body
* Body weight of > 300 lbs. (weight limit of the MRI table)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 45 subjects (male and female) aged 65 and above scheduled for open or laparoscopic general surgical procedures under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2024-05-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative Delirium Incidence | on postoperative day 1
  postoperative delirium will be assessed using 3-Minute Diagnostic Interview for Confusion Assessment Method (CAM)
Postoperative Cognitive Decline | one week before the surgery and postoperative day 7
  postoperative cognitive dysfunction will be assessed using the Montreal Cognitive Assessment (MoCA)
Intraoperative Burst Suppression Time | during the surgical procedure under general anesthesia
  we will use the EEG data recorded during the surgical procedure to calculate time spent in burst suppression

CONTACTS AND LOCATIONS:
Overall Officials: Patrick L. Purdon, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akeju O, Westover MB, Pavone KJ, Sampson AL, Hartnack KE, Brown EN, Purdon PL. Effects of sevoflurane and propofol on frontal electroencephalogram power and coherence. Anesthesiology. 2014 Nov;121(5):990-8. doi: 10.1097/ALN.0000000000000436. PMID 25233374
- [Background] Fournier A, Krause R, Winterer G, Schneider R. Biomarkers of postoperative delirium and cognitive dysfunction. Front Aging Neurosci. 2015 Jun 9;7:112. doi: 10.3389/fnagi.2015.00112. eCollection 2015. PMID 26106326
- [Background] Avidan MS, Fritz BA, Maybrier HR, Muench MR, Escallier KE, Chen Y, Ben Abdallah A, Veselis RA, Hudetz JA, Pagel PS, Noh G, Pryor K, Kaiser H, Arya VK, Pong R, Jacobsohn E, Grocott HP, Choi S, Downey RJ, Inouye SK, Mashour GA. The Prevention of Delirium and Complications Associated with Surgical Treatments (PODCAST) study: protocol for an international multicentre randomised controlled trial. BMJ Open. 2014 Sep 17;4(9):e005651. doi: 10.1136/bmjopen-2014-005651. PMID 25231491
- [Background] Avidan MS, Jacobsohn E, Glick D, Burnside BA, Zhang L, Villafranca A, Karl L, Kamal S, Torres B, O'Connor M, Evers AS, Gradwohl S, Lin N, Palanca BJ, Mashour GA; BAG-RECALL Research Group. Prevention of intraoperative awareness in a high-risk surgical population. N Engl J Med. 2011 Aug 18;365(7):591-600. doi: 10.1056/NEJMoa1100403. PMID 21848460
- [Background] BEDFORD PD. Adverse cerebral effects of anaesthesia on old people. Lancet. 1955 Aug 6;269(6884):259-63. doi: 10.1016/s0140-6736(55)92689-1. No abstract available. PMID 13243706
- [Background] Bennett C, Voss LJ, Barnard JP, Sleigh JW. Practical use of the raw electroencephalogram waveform during general anesthesia: the art and science. Anesth Analg. 2009 Aug;109(2):539-50. doi: 10.1213/ane.0b013e3181a9fc38. PMID 19608830
- [Background] Besch G, Liu N, Samain E, Pericard C, Boichut N, Mercier M, Chazot T, Pili-Floury S. Occurrence of and risk factors for electroencephalogram burst suppression during propofol-remifentanil anaesthesia. Br J Anaesth. 2011 Nov;107(5):749-56. doi: 10.1093/bja/aer235. Epub 2011 Aug 8. PMID 21828343
- [Background] Brice DD, Hetherington RR, Utting JE. A simple study of awareness and dreaming during anaesthesia. Br J Anaesth. 1970 Jun;42(6):535-42. doi: 10.1093/bja/42.6.535. No abstract available. PMID 5423844
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Bruhn J, Bouillon TW, Shafer SL. Bispectral index (BIS) and burst suppression: revealing a part of the BIS algorithm. J Clin Monit Comput. 2000;16(8):593-6. doi: 10.1023/A:1012216600170. PMID 12580235
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Chemali J, Ching S, Purdon PL, Solt K, Brown EN. Burst suppression probability algorithms: state-space methods for tracking EEG burst suppression. J Neural Eng. 2013 Oct;10(5):056017. doi: 10.1088/1741-2560/10/5/056017. Epub 2013 Sep 10. PMID 24018288
- [Background] Ching S, Cimenser A, Purdon PL, Brown EN, Kopell NJ. Thalamocortical model for a propofol-induced alpha-rhythm associated with loss of consciousness. Proc Natl Acad Sci U S A. 2010 Dec 28;107(52):22665-70. doi: 10.1073/pnas.1017069108. Epub 2010 Dec 13. PMID 21149695
- [Background] Flores FJ, Hartnack KE, Fath AB, Kim SE, Wilson MA, Brown EN, Purdon PL. Thalamocortical synchronization during induction and emergence from propofol-induced unconsciousness. Proc Natl Acad Sci U S A. 2017 Aug 8;114(32):E6660-E6668. doi: 10.1073/pnas.1700148114. Epub 2017 Jul 25. PMID 28743752
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Guidera JA, Taylor NE, Lee JT, Vlasov KY, Pei J, Stephen EP, Mayo JP, Brown EN, Solt K. Sevoflurane Induces Coherent Slow-Delta Oscillations in Rats. Front Neural Circuits. 2017 Jul 4;11:36. doi: 10.3389/fncir.2017.00036. eCollection 2017. PMID 28725184
- [Background] Hussain M, Berger M, Eckenhoff RG, Seitz DP. General anesthetic and the risk of dementia in elderly patients: current insights. Clin Interv Aging. 2014 Sep 24;9:1619-28. doi: 10.2147/CIA.S49680. eCollection 2014. PMID 25284995
- [Background] Iwakiri H, Nishihara N, Nagata O, Matsukawa T, Ozaki M, Sessler DI. Individual effect-site concentrations of propofol are similar at loss of consciousness and at awakening. Anesth Analg. 2005 Jan;100(1):107-110. doi: 10.1213/01.ANE.0000139358.15909.EA. PMID 15616062
- [Background] Krenk L, Rasmussen LS. Postoperative delirium and postoperative cognitive dysfunction in the elderly - what are the differences? Minerva Anestesiol. 2011 Jul;77(7):742-9. PMID 21709661
- [Background] Lewis LD, Ching S, Weiner VS, Peterfreund RA, Eskandar EN, Cash SS, Brown EN, Purdon PL. Local cortical dynamics of burst suppression in the anaesthetized brain. Brain. 2013 Sep;136(Pt 9):2727-37. doi: 10.1093/brain/awt174. Epub 2013 Jul 25. PMID 23887187
- [Background] Lewis LD, Weiner VS, Mukamel EA, Donoghue JA, Eskandar EN, Madsen JR, Anderson WS, Hochberg LR, Cash SS, Brown EN, Purdon PL. Rapid fragmentation of neuronal networks at the onset of propofol-induced unconsciousness. Proc Natl Acad Sci U S A. 2012 Dec 4;109(49):E3377-86. doi: 10.1073/pnas.1210907109. Epub 2012 Nov 5. PMID 23129622
- [Background] Mapleson WW. Effect of age on MAC in humans: a meta-analysis. Br J Anaesth. 1996 Feb;76(2):179-85. doi: 10.1093/bja/76.2.179. PMID 8777094
- [Background] Marcantonio ER, Ngo LH, O'Connor M, Jones RN, Crane PK, Metzger ED, Inouye SK. 3D-CAM: derivation and validation of a 3-minute diagnostic interview for CAM-defined delirium: a cross-sectional diagnostic test study. Ann Intern Med. 2014 Oct 21;161(8):554-61. doi: 10.7326/M14-0865. PMID 25329203
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Purdon PL, Pavone KJ, Akeju O, Smith AC, Sampson AL, Lee J, Zhou DW, Solt K, Brown EN. The Ageing Brain: Age-dependent changes in the electroencephalogram during propofol and sevoflurane general anaesthesia. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i46-i57. doi: 10.1093/bja/aev213. PMID 26174300
- [Background] Purdon PL, Pierce ET, Mukamel EA, Prerau MJ, Walsh JL, Wong KF, Salazar-Gomez AF, Harrell PG, Sampson AL, Cimenser A, Ching S, Kopell NJ, Tavares-Stoeckel C, Habeeb K, Merhar R, Brown EN. Electroencephalogram signatures of loss and recovery of consciousness from propofol. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):E1142-51. doi: 10.1073/pnas.1221180110. Epub 2013 Mar 4. PMID 23487781
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Radtke FM, Franck M, Lendner J, Kruger S, Wernecke KD, Spies CD. Monitoring depth of anaesthesia in a randomized trial decreases the rate of postoperative delirium but not postoperative cognitive dysfunction. Br J Anaesth. 2013 Jun;110 Suppl 1:i98-105. doi: 10.1093/bja/aet055. Epub 2013 Mar 28. PMID 23539235
- [Background] Rundshagen I. Postoperative cognitive dysfunction. Dtsch Arztebl Int. 2014 Feb 21;111(8):119-25. doi: 10.3238/arztebl.2014.0119. PMID 24622758
- [Background] Schnider TW, Minto CF, Shafer SL, Gambus PL, Andresen C, Goodale DB, Youngs EJ. The influence of age on propofol pharmacodynamics. Anesthesiology. 1999 Jun;90(6):1502-16. doi: 10.1097/00000542-199906000-00003. PMID 10360845
- [Background] Sebel PS, Bowdle TA, Ghoneim MM, Rampil IJ, Padilla RE, Gan TJ, Domino KB. The incidence of awareness during anesthesia: a multicenter United States study. Anesth Analg. 2004 Sep;99(3):833-839. doi: 10.1213/01.ANE.0000130261.90896.6C. PMID 15333419
- [Background] Soehle M, Dittmann A, Ellerkmann RK, Baumgarten G, Putensen C, Guenther U. Intraoperative burst suppression is associated with postoperative delirium following cardiac surgery: a prospective, observational study. BMC Anesthesiol. 2015 Apr 28;15:61. doi: 10.1186/s12871-015-0051-7. PMID 25928189
- [Background] Steinmetz J, Rasmussen LS. Peri-operative cognitive dysfunction and protection. Anaesthesia. 2016 Jan;71 Suppl 1:58-63. doi: 10.1111/anae.13308. PMID 26620148
- [Background] Strom C, Rasmussen LS, Sieber FE. Should general anaesthesia be avoided in the elderly? Anaesthesia. 2014 Jan;69 Suppl 1(Suppl 1):35-44. doi: 10.1111/anae.12493. PMID 24303859
- [Background] Vutskits L, Xie Z. Lasting impact of general anaesthesia on the brain: mechanisms and relevance. Nat Rev Neurosci. 2016 Oct 18;17(11):705-717. doi: 10.1038/nrn.2016.128. PMID 27752068